CLINICAL TRIAL: NCT06032182
Title: PSYCHE Cognitive Remediation & Social Recovery in Early Psychosis Study
Brief Title: PSYCHE Cognitive Remediation & Social Recovery Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Service Executive, Ireland (Other); Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Gary Donohoe, Professor Gary Donohoe, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUIRELAND2
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Early Psychosis
Keywords: Recovery; Cognitive remediation training; Cognitive behavioural therapy; Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 15 sessions of the combined cognitive remediation training and social recovery therapy intervention.
  Interventions: Behavioral: CRESTR Intervention
- Control (Active Comparator): 15 sessions of social recovery therapy alone.
  Interventions: Behavioral: CRESTR Control

INTERVENTIONS:
Behavioral: CRESTR Intervention — 15 1-hour sessions of CRT + SRT
  Arms: Intervention
Behavioral: CRESTR Control — 15 1-hour sessions of SRT alone
  Arms: Control

SUMMARY:
This study is a pilot feasibility study embedded in the Early Intervention in Psychosis (EIP) services in Ireland. It explores the feasibility and acceptability of a combined cognitive remediation training and social recovery therapy intervention.

DETAILED DESCRIPTION:
The Cognitive Remediation and Social Recovery in Early Psychosis (CRESTR) study is a feasibility study recruiting participants from the Health Service Executive Early Intervention in Psychosis (EIP) services in Sligo, Meath and Cork and the Adult Mental Heath Service in Galway. This study explores the feasibility and acceptability of a novel, 15-week multicomponent psychosocial intervention which combines cognitive remediation training (CRT) and social recovery therapy (SRT). Primary and secondary outcome measures are described later in this registration. The intervention components include:

Component 1: The CRT programme used in this study is the Computerised Interactive Remediation of Cognition- Training for Schizophrenia (CIRCuiTS). CIRCuiTS is a web-based CRT programme which targets metacognition, specifically strategy use, in addition to massed practice of cognitive functions (attention, memory and executive functioning). Collaborative goal setting related to real-world tasks are integral to the programme with the programme tasks and exercises increasing in difficulty in response to the participant's performance and progress. This will be the primary focus of 1:1 therapy for the first 7 weeks with remote practice sessions occurring between therapy visits. After 7 weeks remote practice will continue and the focus of in-person therapy sessions will bridge to social recovery therapy as detailed below.

Component 2: Social recovery therapy (SRT) focuses on addressing barriers to individuals interacting in their social environment e.g., social anxiety. It is informed by cognitive behavioural theory and addresses individual goals. SRT follows an established protocol. In summary, this consists of therapy delivered in three stages. Stage one will include engagement and formulation with the purpose of identifying a problem list and establishing a therapeutic relationship. Stage two will include preparing for new activities with identification of pathways to activity and collaboration with community stakeholders. Stage three will include engagement in new activities using behavioural experiments to promote social activity. This is the primary focus of in-person therapy sessions from week 8 to 15 alongside remote practice of the CRT programme.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years of age
* Within the first 5 years of a diagnosed psychotic disorder
* Community based and clinically stable
* Ability to give informed consent

Exclusion Criteria:

* History of organic impairment
* IQ< 70
* History of head injury with loss of consciousness > 5-minute duration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Social and Occupational Functioning Assessment Scale | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  Social and Occupational Functional Assessment Scale (Rybarczyk, 2011) is a global rating of current functioning ranging from 0 to 100, with lower scores representing lower functioning.

SECONDARY OUTCOMES:
The Reading the Mind in the Eyes Task | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Reading the mind in the eyes task is a theory of mind task that measures the capacity to understand mental states of others from expressions in the eye region of the face. Participants view 36 photos and choose the most accurate descriptor word from four choices for the thought/feeling that was portrayed. Scores range from 0 to 36 with higher scores indicating better theory of mind ability.
Emotion Recognition Task | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Emotion Recognition Task from the Cambridge Neuropsychological Test Automated Battery (Cambridge Cognition Ltd.)
  Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise).
  The outcome measures for ERT will include number correct, which can be looked at either across individual emotions or across all emotions at once. Higher scores indicate superior emotion recognition ability.
The Bell Lysaker Emotion Recognition Task | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Bell Lysaker Emotion Recognition Task measures recognition of seven emotional states: happiness, sadness, fear, disgust, surprise, anger, or no emotion. Participants identified the emotion shown in 21 videos of a male actor providing dynamic facial, vocal-tonal, and upper-body movement cues. Performance is indexed as the total number of correctly identified emotions (ranging from 0 to 21 i.e. a higher score represents superior emotion recognition ability.
Test of Premorbid Functioning | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  Test of Premorbid Functioning estimates an individual's pre-morbid cognitive and memory functioning. A revised and updated version of the Wechsler Test of Adult Reading™, TOPF helps predict pre-injury IQ and memory abilities. Total score is derived from the number of correct items, ranges from 0-70 with a higher score indicating superior ability.
The matrix reasoning subtest from the Wechsler Adult Scale of Intelligence 3rd edition (WAIS-III) | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The matrix reasoning subtest from the Wechsler Adult Scale of Intelligence 3rd edition (WAIS-III) (Wechsler, 1997) is a brief, reliable measure of cognitive ability for use in clinical, educational and research settings. Matrix reasoning subtest scores range from 0 - 26 with higher scores reflecting better perceptual organization. Once raw scores are derived they are converted to scaled scores adjusted for age.
Letter Number Sequencing Task | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The letter-number sequencing task from the Wechsler Memory scale 3rd edition WMS-III assesses working memory. Scores range from 0-21. Higher scores on the WMS-III subtests indicate better memory function. Raw scores are converted to scaled scores adjusted for age.
Metacognitive Awareness Scale, Domain Specific | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  Meta-Cognitive Awareness Scale - Domain Specific encourages reflection of task strategy processes. This domain-specific scale was first constructed to measure participants' awareness of their own metacognition linked to Raven's Progressive Matrices (SPM). Following discriminatory index and Exploratory Factor Analysis, a 15-item scale was derived. Exploratory Factor Analysis showed five factors: Awareness of Engagement in Self-Monitoring, Awareness of Own Ability, Awareness of Responding Speed/Time, Awareness of Alternative Solutions and Awareness of Requisite Problem-Solving Resources. The total score is the sum of the 15-itm scale with higher scores indicating superior metacognitive awareness.
The Scale for the Assessment of Positive Symptoms and the Scale for the Assessment of Negative Symptoms. | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Scale for the Assessment of Positive Symptoms measures positive symptoms on a 24 item scale, this includes 19 negative symptom item ratings, and 5 global factor ratings. Each item is scored on a six point scale from 0-5. The composite total is the sum of the nineteen item ratings. The SANS global total is the sum of the five global ratings. The higher the score the more symptomology or severity of symptoms.
  The Scale for the Assessment of Negative Symptoms measures negative symptoms on a 25 item, 6-point scale from 0-5. Items are listed under the five domains of affective blunting, alogia, avolition/apathy, anhedonia/asociality, and attention. Total (Composite) score is calculated as the sum of SANS items 1-7, 9-12, 14-16, 18-21, and 23-24, while SANS (Global) Summary score was calculated as the sum of SANS items 8, 13, 17, 22, and 25. The higher the score the more symptomology or severity of symptoms.
The Patient Health Questionnaire-9 | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Patient Health Questionnaire-9 is a brief tool used to diagnose and measure severity of depression. It is adapted from the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV). Scores range from 0 to 27 with higher scores indicating more severe depression.
  A total score of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
The Generalised Anxiety Disorder Assessment-7 | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Generalised Anxiety Disorder Assessment is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Total scores range from 0 to 21with higher scores indicating a higher level of anxiety. Clinical categorisations of anxiety levels are: 0-4 (none), 5-9 (mild), 10-14 (moderate), and 15-21 (severe).
Drug Use Disorders Identification Test | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Drug Use Disorders Identification Test is an 11-item self-administered screening instrument for drug-related problems, giving information on the level of drug intake and selected criteria for substance abuse/harmful use and dependence according to the ICD-10 and DSM-4 diagnostic systems. The minimum total score possible is 0, and the maximum total score possible is 44 (i.e. total score range: 0-44). Higher scores reflect higher drug dependence
Alcohol Use Disorders Identification Test | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Alcohol Use Disorders Identification Test is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviors, and alcohol-related problems. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption according to World Health Organization (WHO) guidelines. Scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
EQ-ED-EL Health Questionnaire | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on scale that describes the degree of problems in that area (i.e. I have no problems walking about, slight problems, moderate problems, severe problems, or unable to walk). This tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.
Global Functioning Scale | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Global Functioning Scale: Role: measures performance and amount of support needed in one's specific role (ie, school, work). Social: measures quantity and quality of peer relationships, level of peer conflict, age-appropriate intimate relationships, and involvement with family members. Scale: 1-10, higher scores indicate better functioning.
MIRECC Global Assessment of Function | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The MIRECC Global Assessment of Function measures occupational functioning, social functioning, and symptom severity on 3 subscales. 3 subscales scored from 0 to 100, with higher scores indicating better functioning.
Global Assessment of Function | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Global Assessment of Function scale is a 100-point single-item scale designed to measure the global severity of psychiatric illness on the basis of symptom, social, and occupational functioning combined. The scale is divided into 10 anchor intervals, with descriptions and examples of symptoms and of social and occupational functioning. Higher scores indicate better functioning.
Time Use Survey | T0 (Baseline) T1 (1-2 weeks post intervention) T2 (3-month follow up)
  The Time Use Survey is a semi-structured interview that enquires about time spent over the past month on work, education, voluntary work, leisure, sports, housework or chores, and child care. Time spent on each of the activities is calculated in terms of the average number of hours per week. The activities are summed to create two scores: constructive economic activity (work, education, voluntary work, housework or chores, and child care) and structured activity (constructive economic activity plus leisure and sports activities). Less than 45 hours of structured activity per week is considered a threshold for being at risk of social disability, less than 30 hours per week is threshold for social disability and indicative of poor social functioning, and less than 15 hours per week is considered to reflect serious social disability.

CONTACTS AND LOCATIONS:
Locations (5):
- Ireland (5):
  - HSE Early Intervention in Psychosis Service, Cork, Cork
  - DETECT Early Intervention in Psychosis Service, Dublin
  - Adult Mental Health Service, University Hospital Galway, Galway
  - HSE Early Intervention in Psychosis Service, Meath, Navan
  - HSE Early Intervention in Psychosis Service, Sligo, Sligo

IPD SHARING:
Plan to Share IPD: Yes
The full protocol in addition to datasets and statistical code generated during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: The full protocol in addition to datasets and statistical code generated during the current study will be available from the corresponding author on reasonable request.